CLINICAL TRIAL: NCT00335335
Title: Phase 3, Open-label, Multicenter Studies to Determine Efficacy and Safety of VISIPAQUETM (Iodixanol) Injection for Use in Intravenous Contrast-Enhanced CT Angiography of Coronary Arteries
Brief Title: Safety and Effectiveness of Visipaque 320mg-I/ml for Use in Contrast-Enhanced CT Angiography of Arteries of the Heart
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision due to low subject recrcuitment
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DXV301
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary; Angiography; X-ray; CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — iodixanol

ARMS (1):
- Visipaque Injection (Experimental): All participants will receive intravenous (IV) administration of 80 mL Visipaque (iodixanol) 320 mg-I/mL at a rate of 4-5 mL per second via power injector followed by a saline injection of 40-50 mL 0.9% sodium chloride solution at a rate of 4-5 mL per second.
  Interventions: Drug: iodixanol

INTERVENTIONS:
Drug: iodixanol
  Other Names: Visipaque

SUMMARY:
CT (computed tomography) angiography (CTA) is an examination similar to a CAT scan that uses x-rays and a contrast medium (also called dye) to visualize blood flow in arteries and veins throughout the body.

VISIPAQUE™ will be given through a vein in the arm before having the CTA scan of the heart arteries. The pictures it produces of the heart and its blood vessels will be reviewed and compared to those obtained during the catheter-based coronary angiography to see if the CTA shows the same blockages.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years old.
* Subject must have been referred for an elective coronary angiography for one of several specified conditions.

Exclusion Criteria:

* The subject has impaired renal function with a serum creatinine level ≥1.7 mg/dL (150 µmol/L). If the institution's practising guideline(s) regarding the serum creatinine limits for receiving radiologic contrast medium are lower than 1.7 mg/dL (150 µmol/L), the investigator should follow the practising guideline(s) of their institution.

Subject has a known allergy to iodinated contrast agent

Subject has atrial fibrillation/flutter or any irregular heart rhythm considered to interfere with temporal acquisition of cardiac CT images.

The subject's resting heart rate is 66-100 bpm and β-blocker therapy is contraindicated.

Use of nitroglycerin is contraindicated.

Subject has had a prior CABG procedure.

Subject has a metal cardiac stent in place or artificial heart valve(s).

Subject has had a prior pacemaker or internal defibrillator lead implantation. Subject must agree to discontinue metformin day of and for 48 hours after the CTA procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12-02 (Actual); Study Completion 2006-12-02 (Actual)

PRIMARY OUTCOMES:
To evaluate diagnostic performance and safety of Visipaque-enhanced CTA images for determination of presence or absence of coronary artery obstruction | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Reichl, Study Director — GE Healthcare
Locations (1):
- Princeton, New Jersey, United States